CLINICAL TRIAL: NCT01066611
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Two-Period Crossover Study to Investigate the Safety of CAL-263 in Allergic Rhinitis Subjects and Effects on the Response to Environmental Chamber Allergen Challenge
Brief Title: Study to Investigate Effects of CAL-263 in Subjects With Allergic Rhinitis Exposed to Allergen in an Environmental Chamber
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Langdon Miller, M.D., VP Clinical Research, Oncology, Gilead Sciences
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 263-02
Record Dates: First submitted 2010-01-27; First posted 2010-02-10 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Allergy; Phosphatidylinositol 3-kinase
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): CAL-263
  Interventions: Drug: CAL-263
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CAL-263 — CAL-263 10 mg or placebo once daily for 7 days
  Arms: 1
Drug: Placebo — CAL-263 10 mg or placebo once daily for 7 days
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety and effect of CAL-263 in subjects with allergic rhinitis.

DETAILED DESCRIPTION:
A Phase I, randomized, double-blind crossover study of CAL-263, an oral inhibitor of PI3K delta, in patients with allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 and <55 years
2. Has a history of seasonal allergic rhinitis for at least 2 years
3. Has sensitivity to grass pollen demonstrated by a positive response to skin prick testing
4. Has a positive Radio Allergen Sorbent Test (class 2 or greater) for grass pollen during the previous 12 months or at screening
5. Is otherwise healthy
6. Is able to provide written informed consent

Exclusion Criteria:

1. Is a female of childbearing
2. History of chronic nasal or upper respiratory tract symptoms or disorders other than allergic rhinitis
3. History of nonallergic rhinitis, chronic sinusitis or severe asthma
4. Has a nasal condition likely to affect the outcome of the study
5. Is currently taking regular medication, whether prescribed or not, including corticosteroids, vitamins, macrolides, anti-fungal agents and herbal remedies
6. Has taken a prohibited medication within the specified interval prior to Visit 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of CAL-263 in allergic rhinitis subjects | 46 days

SECONDARY OUTCOMES:
Determine the efficacy of CAL-263 on total nasal symptom scores following an allergen challenge in allergic rhinitis subjects | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Horak, MD, Principal Investigator — Vienna Challenge Chamber
Locations (1):
- Vienna Challenge Chamber, Vienna, Austria